CLINICAL TRIAL: NCT02535871
Title: A Phase 3, Multi-Center, Randomized, Double-Blind, Vehicle-Controlled, 2-Arm, Parallel Group Comparison Study Comparing the Efficacy and Safety of IDP-121 and IDP-121 Vehicle Lotion in the Treatment of Acne Vulgaris
Brief Title: A Study Comparing the Efficacy and Safety of IDP-121 and IDP-121 Vehicle Lotion in the Treatment of Acne Vulgaris
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Valeant Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: V01-121A-302
Record Dates: First submitted 2015-08-26; First posted 2015-08-31 (Estimated); Last update posted 2015-09-14 (Estimated); Status verified 2015-09

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDP-121 Lotion (Experimental): IDP-121 Lotion, applied topically to the face, once daily for 12 weeks.
  Interventions: Drug: IDP-121 Lotion
- IDP-121 Lotion Vehicle (Placebo Comparator): IDP-121 Vehicle Lotion, applied topically to the face, once daily for 12 weeks
  Interventions: Drug: IDP-121 Vehicle Lotion

INTERVENTIONS:
Drug: IDP-121 Lotion — Investigational Product: IDP-121 Lotion
  Arms: IDP-121 Lotion
Drug: IDP-121 Vehicle Lotion — Comparator Product: IDP-121 Vehicle Lotion
  Arms: IDP-121 Lotion Vehicle

SUMMARY:
The primary objective of this study is to compare the efficacy, safety and tolerability of IDP-121 Lotion and vehicle in the treatment of subjects with acne vulgaris.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, parallel group, vehicle-controlled, 12-week study to evaluate relative changes in inflammatory and non-inflammatory lesion counts, as well as treatment success using an Evaluator's Global Severity Scale (EGSS) in subjects with moderate to severe acne. IDP-121 is a lotion for the topical treatment of acne.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 9 years of age and older
* Written and verbal informed consent must be obtained.
* Subject must have a score moderate or severe on the Evaluator's Global Severity assessment at the screening and baseline visit
* Pre-menses females and women of childbearing potential must have a negative urine pregnancy test at the screening and baseline visits
* Subjects must be willing to comply with study instructions and return to the clinic for required visits.

Exclusion Criteria:

* Any dermatological conditions on the face that could interfere with clinical evaluations
* Any underlying disease(s) or some other dermatological condition of the face that requires the use of interfering topical or systemic therapy or makes evaluations and lesion count inconclusive
* Subjects with a facial beard or mustache that could interfere with the study assessments
* Concomitant use of potentially irritating over-the-counter products

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Absolute change in inflammatory lesion count from baseline to Week 12 | 12 weeks
  At each visit the Evaluator will count the total number of inflammatory lesions (papules, pustules, and nodules) on the subject's face.
  Inflammatory lesions are defined as follows:
  Papule - a small, solid elevation less than 5 mm in diameter. Most of the lesion is above the surface of the skin.
  Pustule - a small, circumscribed elevation less than 5 mm in diameter that contains yellow-white exudate.
  Nodule - a subcutaneous lesion greater than or equal to 5 mm in diameter.
Absolute change in non-inflammatory lesion count from baseline to Week 12 | 12 weeks
  At each visit the Evaluator will count the total number of non-inflammatory lesions (open and closed comedones).
  Non-inflammatory lesions are defined as follows:
  Open comedones (black head) - a lesion in which the follicle opening is widely dilated with the contents protruding out onto the surface of the skin.
  Closed comedones (white head)- a lesion in which the follicle opening is closed, but the sebaceous gland is enlarged by the pressure of the sebum build up, which in turn causes the skin around the follicle to thin and become elevated with a white appearance.
Proportion of subjects who have a least a 2 grade reduction at Week 12 from baseline in the Evaluator's Global Severity Score and were Clear or Almost Clear | 12 weeks
  At each visit the severity will be determined based on evaluator-blinded evaluations of the signs and symptoms of acne vulgaris. Evaluations will be scored on a scale of 0-4 (Evaluator's Global Severity Score), with 0 being clear and 4 being severe. Please see below for complete definitions.
  0 - Clear - Normal, clear skin with no evidence of acne vulgaris
  1. Almost clear- Rare non-inflammatory lesions present, with rare non-inflamed papules (papules must be resolving and may be hyperpigmented, though not pink-red)
  2. Mild- Some non-inflammatory lesions are present, with few inflammatory lesions (papules/pustules only; no nodulo-cystic lesions)
  3. Moderate-Non-inflammatory lesions predominate, with multiple inflammatory lesions evident: several to many comedones and papules/pustules, and there may or may not be one nodulo-cystic lesion
  4. Severe- Inflammatory lesions are more apparent, many comedones and papules/pustules, there may or may not be up to 2 nodulo-cystic lesions.

SECONDARY OUTCOMES:
Percent change in inflammatory lesion count from baseline to Week 4, 8, and 12 | 4, 8, and 12 weeks
  At each visit the Evaluator will count the total number of inflammatory lesions (papules, pustules, and nodules) on the subject's face, and the percent change will be calculated.
Percent change in non-inflammatory lesion count from baseline to Week 4, 8, and 12 | 4, 8, and 12 weeks
  At each visit the Evaluator will count the total number of non-inflammatory lesions (open and closed comedones), and the percent change will be calculated.
Proportion of subjects who have a least a 2 grade reduction at Week 4, 8, and 12 from baseline in the Evaluator's Global Severity Score | 4, 8, and 12 weeks
  At each visit the severity will be determined based on evaluator-blinded evaluations of the signs and symptoms of acne vulgaris. Evaluations will be scored on a scale of 0-4 (Evaluator's Global Severity Score), with 0 being clear and 4 being severe. Please see below for complete definitions.
  0 - Clear - Normal, clear skin with no evidence of acne vulgaris
  1. Almost clear- Rare non-inflammatory lesions present, with rare non-inflamed papules (papules must be resolving and may be hyperpigmented, though not pink-red)
  2. Mild- Some non-inflammatory lesions are present, with few inflammatory lesions (papules/pustules only; no nodulo-cystic lesions)
  3. Moderate-Non-inflammatory lesions predominate, with multiple inflammatory lesions evident: several to many comedones and papules/pustules, and there may or may not be one nodulo-cystic lesion
  4. Severe- Inflammatory lesions are more apparent, many comedones and papules/pustules, there may or may not be up to 2 nodulo-cystic lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Anya Loncaric, MS, Study Director — Valeant Pharmaceuticals